CLINICAL TRIAL: NCT03466125
Title: Massachusetts-wide Study of the Incidence of ATrial Fibrillation and Stroke Occurring After Discharge From Cardiac Surgery (MATRICeS)
Brief Title: Characterization and Prediction of Atrial Fibrillation-caused Adverse Events After Hospital Discharge for Cardiac Surgery
Acronym: MATRICeS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Baystate Medical Center (Other); Cape Cod Hospital (Other); Mount Auburn Hospital (Other); Memorial University Medical Center (Other); Tufts Medical Center (Other); St. Elizabeth's Medical Center (Unknown); SouthCoast Medical Group (Other)
Responsible Party: Principal Investigator, Jochen Daniel Muehlschlegel, MD, Vice Chair of Research, Brigham and Women's Hospital
Other Study IDs: 2017P002261
Record Dates: First submitted 2018-03-05; First posted 2018-03-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Stroke, Acute; Death
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Death | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients who underwent cardiac surgery in Massachusetts: No interventions. A retrospective cohort study of patients who underwent cardiac surgery in Massachusetts in calendar years 2012 - 2016.
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Retrospective cohort study

SUMMARY:
The purpose of the research is to identify the frequency and severity of adverse events related to atrial fibrillation that occur after discharge from hospital where the patient underwent cardiac surgery.

The Specific Aims of the proposed study are to:

1. Identify the predictors of postoperative atrial fibrillation after discharge from hospital.
2. Identify the frequency of readmission to hospital, or other resource use such as Emergency Department or outpatient visit, for the treatment or prophylaxis of postoperative AF and consequent stroke or bleeding outcomes.
3. Identify the risks for stroke, death and other morbidity in patients after cardiac surgery and the effect of postoperative AF upon subsequent stroke or bleeding outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cardiac surgery in Massachusetts between 2012 - 2016

Exclusion Criteria:

* surgical procedures that do not include coronary artery bypass graft surgery, aortic valve surgery or mitral valve surgery;
* surgical procedures that include MAZE surgery, or pulmonary vein isolation, ventricular assist device, heart transplantation, congenital heart surgery, bacterial endocarditis, cardiac trauma, cardiac tumor, ventricular septal defect repair, left ventricular aneurysm repair, pulmonary thromboendarterectomy, sub-aortic stenosis resection or surgical ventricular restoration;
* surgical procedures on patients that have undergone MAZE surgery, AF ablation procedures, pulmonary vein isolation or left atrial appendage resection or ablation (such as Watchman devices).

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent cardiac surgery in Massachusetts between 2012 - 2016
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recurrent atrial fibrillation | Up to six years after surgery
  Recurrent atrial fibrillation
Acute ischemic stroke | Up to six years after surgery
  Acute ischemic stroke
Mortality | Up to six years after surgery
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jochen D Muehlschlegel, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03466125/Prot_SAP_000.pdf